CLINICAL TRIAL: NCT06607861
Title: Nebulized Dexmedetomidine or Lidocaine for Treatment of Post Dural Puncture Headache in Parturients Undergoing Elective Cesarean Section Under Spinal Anesthesia: A Randomized Bicentric Study
Brief Title: Nebulized Dexmedetomidine or Lidocaine for Treatment of Post Dural Puncture Headache in Parturients Undergoing Elective Cesarean Section Under Spinal Anesthesia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R/603- Anet19-1
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pain Score (VAS)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): nebulization of 4 mL 0.9% saline plus conventional management ( consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol plus 130 mg caffeine every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: saline group
- Dex. group (Active Comparator): nebulization of 1 µg/kg dexmedetomidine diluted in 4 mL 0.9% saline twice daily ( fixed times 9 a.m, and 9 p.m) plus conventional management ( consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol plus 130 mg caffeine every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: dexmedetomidine group
- Lidocaine group (Active Comparator): bilateral nebulization (60 mg) using a mucosal atomization device twice daily plus conventional management ( consisted of bed rest in the supine position, good hydration with continuous infusion of 30 mL/kg/day lactated Ringer solution, 1 g paracetamol plus 130 mg caffeine every 6 h. Diclofenac sodium suppository (100 mg) was given twice daily for 5 days as routine post-operative pain management
  Interventions: Drug: lidocaine group

INTERVENTIONS:
Drug: saline group — nebulization of 4 mL 0.9% saline twice daily
  Other Names: nebulization of 4 mL 0.9% saline twice daily
  Arms: Control group
Drug: dexmedetomidine group — nebulization of 1 µg/kg dexmedetomidine diluted in 4 mL 0.9% saline twice daily
  Arms: Dex. group
Drug: lidocaine group — bilateral nebulization (60 mg) using a mucosal atomization device twice daily
  Arms: Lidocaine group

SUMMARY:
Post-dural puncture headache (PDPH) is a well-recognized and potentially serious complication of subarachnoid block. While advancements in spinal needle design have reduced its incidence in recent years, PDPH still affects a notable percentage of post-partum patients undergoing spinal anaesthesia, with rates ranging from 0.5% to 2%. Factors such as female gender, pregnancy, young age, low body mass index, dilutional anemia, and the preference for neuraxial anaesthesia during caesarean section (CS) increase the vulnerability of obstetric patients to PDPH. Therefore, managing this complication is critically important in obstetric anaesthesia.

The exact cause of PDPH remains unclear, but there is substantial evidence suggesting that it stems from reduced cerebrospinal fluid (CSF) pressure due to continuous leakage through a dural tear, which exceeds the rate of CSF production. This imbalance can lead to PDPH, as even a modest loss of CSF volume (as little as 10%) can trigger traction on pain-sensitive intracranial structures when in an upright position, compounded by reflexive vasodilation.

Various treatment strategies have been proposed, typically including bed rest in a supine position, fluid therapy, analgesics, and medications such as sumatriptan and caffeine.

Dexmedetomidine (DEX) is a highly specific agonist of α2-adrenoreceptors known for inducing cooperative sedation, anxiolysis, and analgesia while minimizing respiratory depression. Additionally, it has been shown to mitigate the stress and inflammatory response triggered by surgical and anaesthetic procedures. Activation of α2-receptors in the substantia gelatinosa of the dorsal horn suppresses the firing of nociceptive neurons and inhibits the release of substance P. Furthermore, stimulation of these receptors in the locus coeruleus, a key modulator of nociceptive transmission, interrupts the transmission of pain signals, resulting in analgesia. Dexmedetomidine has been administered via intranasal and inhalational routes for various purposes, including premedication, sedation, and post-operative analgesia.

Lidocaine nebulized is a novel method used recently for PDPH. Intranasal lidocaine can offer sphenopalatine ganglion block which can facilitate acute pain reduction in PDPH.

ELIGIBILITY:
Inclusion Criteria:

* Post partum headache for parturient with elective CS under spinal anesthesia with visual analog score (VAS) ≥ 4 [14] and Lybecker classification score ≥ 2

Exclusion Criteria:

* Emergency caesarean section.
* Pregnancy induced hypertension
* Contraindications for sub-arachinoid block ( coagulopathy, infection )
* History of chronic headache, migraine, trigeminal neuralgia
* Refusal to participate
* History of cerebrovascular stroke
* BMI> 35
* History of obstructive sleep apnea.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Pain severity | at enrollment,1,3,6, 12, 24,36, 48, 72 hours
  Visual analogue scale from 0 to ten . 0 = no pain. 1-3=mild pain, 4-6= moderate. 7- 10= severe un imaginable pain

SECONDARY OUTCOMES:
leybecker classification | At enrollment, 1,3,6, 12,24,36,48, 73 hours
  degree of headache ... <2 = mild pain.. > 2= severe pain
Transcranial doppler | at enrollment, 24,48,72 hours
  Measuring mean flow velocity
NEED for epidural blood patch | 72 hours during the invesigation
  Visual analogue scale from 0 to ten . 0 = no pain. 1-3=mild pain, 4-6= moderate. 7- 10= severe un imaginable pain. Epidural blood patch if visual analogue scale more than or equal 4.
Procedural related complications | 72 hours from the procedure
  hypotension, bradycardia
persistent symptoms | one week after hospital discharge
  Tinnitus, photophobia, orthostatic hypotension
transcranial doppler | at enrollment, 24,48,72 hours
  pulsatality index
transcranial doppler | at enrollment, 24,48,72 hours
  resisitive index